CLINICAL TRIAL: NCT06212882
Title: Dual-Energy CT Angiography in Suspected Pulmonary Embolism: Influence of Concentration of Contrast Materials on Image Quality and Diagnostic Performance
Brief Title: Optimization of DE-CTPA Images and Diagnostic Pathway: Using Low Concentration Iodine Contrast Material
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Principal Investigator, Peihua Lu, Director of Scientific Research Department, Wuxi People's Hospital
Other Study IDs: KY23055
Record Dates: First submitted 2023-12-18; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; Computed Tomography; contrast materials
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lower concentration and lower volume contrast agent group
  Interventions: Diagnostic Test: Lower concentration and lower volume contrast agent group
- Lower concentration and normal volume contrast agent group
  Interventions: Diagnostic Test: Lower concentration and lower volume contrast agent group
- Normal concentration and normal volume contrast agent group

INTERVENTIONS:
Diagnostic Test: Lower concentration and lower volume contrast agent group — CT images using lower concentration and lower volume contrast material
  Groups: Lower concentration and lower volume contrast agent group; Lower concentration and normal volume contrast agent group

SUMMARY:
The investigators aimed to compare the image quality and diagnostic performance of DECTPA using lower concentration iodine contrast materials and using normal concentration iodine contrast materials in the evaluation of suspected pulmonary embolism.

DETAILED DESCRIPTION:
All patients met the inclusion and exclusion criteria will be given written informed consensus. The enrolled patients will randomly receive one of the three injection protocols: A: 30mL Iomeprol (Iomeron 300, Bracco Imaging, Milano, Italia) injected at a flow rate of 4mL/s; B: 50mL Iomeprol (Iomeron 300, Bracco Imaging, Milano, Italia) injected at a flow rate of 4mL/s; C: 50mL Ioversol (Ioversol 350, Hengrui, Jiansun, China) injected at a flow rate of 4mL/s. A and B groups are both lower concentration iodine contrast material groups, with different total iodine loads.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Clinical suspicion of pulmonary embolism suggests CTPA examination (Wells score>4 or D-2 polymer elevation)
* Patient's general physical condition tolerates CTPA examination

Exclusion Criteria:

* Allergy to iodine contrast agents
* Hyperthyroidism
* Pregnancy
* Weight greater than 80kg
* Heart failure patients, NYHA heart function level III or IV

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will undergo CT pulmonary angiography due to clinical suspicion of pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
image quality evaluation of the CTPA images of 30% participants | through the CTPA examinations of 30% participants finished,, an average of six month
  1. the mean CT number (in Hounsfield units) in the main pulmonary artery by using a region of interest of at least 1 square centimeter.
  2. the CT number (in Hounsfield units) of peripheral pulmonary arteries close to the beginning and the end of each scan in a egmental or subsegmental artery at an apical and a basal section position. Because the caliber of the peripheral vessels was too small to reliably set an intraluminal region of interest to determine the mean CT number, the maximum CT number as a proxy for vascular attenuation should be chosen.
  3. the images quality score for making a diagnosis other than PE ( using a five-point scale ranging from 1 to 5).

SECONDARY OUTCOMES:
overall diagnostic performance for pulmonary embolism | CTPA examinations all participants are finished, an average of two month
  diagnostic accuracy, sensitivity and specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
index that measuring image quality and pulmonary embolism CTPA diagnostic results for each individual
Supporting Information: Study Protocol
Time Frame: After the main paper is published.
Access Criteria: application from the Central Contact Person